CLINICAL TRIAL: NCT03944733
Title: Iron Status, Maternal Depressive Symptoms, and Mother-child Interactions
Acronym: IDinteract
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was never started as a result of change of personnel and funding
Sponsor: Penn State University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 00009190
Record Dates: First submitted 2019-04-04; First posted 2019-05-09 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Iron Deficiency Anemia
Keywords: iron deficiency anemia (IDA); iron status; mother-infant interactions; intervention study; postpartum depressive symptoms
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Iron; Gelatin

STUDY DESIGN:
Intervention Model Description: Iron deficient anemic (IDA) mothers will be given an iron supplement versus iron sufficient (control; CN) mothers will be given a placebo (gelatin pill) daily.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A study staff not involved with data analyses or outcome assessment will provide the intervention to participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iron Intervention (Active Comparator): IDA mothers will receive a 65 mg of iron (ferrous sulfate) daily for 4.5 months in the postpartum period (6 weeks to 6 months post delivery).
  Interventions: Dietary Supplement: Iron
- Placebo (Placebo Comparator): IS mothers will receive 600 mg of gelatin daily for 4.5 months in the postpartum period (6 weeks to 6 months post delivery).
  Interventions: Dietary Supplement: Gelatin

INTERVENTIONS:
Dietary Supplement: Iron — 65 mg of iron (ferrous sulfate)
  Other Names: Iron, Spring Valley
  Arms: Iron Intervention
Dietary Supplement: Gelatin — 600 mg gelatin
  Other Names: 21st Century
  Arms: Placebo

SUMMARY:
This study aims to examine the relation between iron status and maternal-child interactions as well as maternal depressive symptoms in mothers from central Pennsylvania.

DETAILED DESCRIPTION:
Investigators aim to follow mothers and their infants from 6 weeks to 6 months in the postpartum to understand the relation between iron status and mother-child interactions and depressive symptoms. During this period, iron deficient anemic mothers will receive an intervention with iron with the scope of improving iron status, reducing their depressive symptoms, and in turn, increasing the quality of parenting behaviors during mother-child interactions. The control group will be iron sufficient mothers who will receive a placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women between 18 - 40 years.
2. Mother expects to be the primary caregiver for the infant for study duration and will allow infant to be enrolled in the study..
3. Mother has no history of gastrointestinal or hematological disorders and not taking medications that interfere with hematopoiesis or absorption.
4. After birth, the mother and baby are healthy, delivery was of one infant only, infant gestational age ≥ 38 weeks, infant weight ≥ 2500 g (5.5 lbs), neither the mom nor the infant received a blood transfusion at or since delivery, and mom agrees to discontinue use of any iron containing medications.

Exclusion Criteria:

1. Maternal age ≤ 18 and > 40 years
2. Evidence of a history of gastrointestinal or hematological disorders and evidence of taking medications that interfere with hematopoiesis or absorption.
3. Severely anemic (Hemoglobin < 90 g/L)
4. Iron deficient but not anemic women
5. Non-English speaking

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Mother-child interaction scores in the postpartum period | 1 year
  Mother child-interactions will be measured via the Emotional Availability Scales and microanalytic coding. Scores will be compared between iron deficient and iron sufficient women. Investigators will also examine change in scores within group from baseline to endline.
  The Emotional Availability Scales consist of 6 subscales, 4 for the mother and 2 for the child. Maternal subscales include sensitivity, structuring, non-intrusiveness, and non-hostility; child subscales include involvement and responsiveness. All are scored on a scale of 1 - 7 with higher scores indicating a more optimal score.

CONTACTS AND LOCATIONS:
Overall Officials: Laura E Murray-Kolb, PhD, Principal Investigator — Penn State University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murray-Kolb LE, Beard JL. Iron deficiency and child and maternal health. Am J Clin Nutr. 2009 Mar;89(3):946S-950S. doi: 10.3945/ajcn.2008.26692D. Epub 2009 Jan 21. PMID 19158210
- [Background] Armony-Sivan R, Kaplan-Estrin M, Jacobson SW, Lozoff B. Iron-deficiency anemia in infancy and mother-infant interaction during feeding. J Dev Behav Pediatr. 2010 May;31(4):326-32. doi: 10.1097/DBP.0b013e3181dc525d. PMID 20431398
- [Background] Corapci F, Radan AE, Lozoff B. Iron deficiency in infancy and mother-child interaction at 5 years. J Dev Behav Pediatr. 2006 Oct;27(5):371-8. doi: 10.1097/00004703-200610000-00001. PMID 17041272